CLINICAL TRIAL: NCT06656936
Title: Expanding Access to Colorectal Cancer Screening Through Community Pharmacies: The PharmFIT Study
Brief Title: The PharmFIT Study
Acronym: PharmFIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LCCC2430; 1R01CA279010-01A1 (NIH)
Record Dates: First submitted 2024-09-16; First posted 2024-10-24 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: Cancer Screening; Colorectal Cancer; Implementation Science; Rural Health; Minority Health; Community Pharmacies
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two or more groups in parallel for the duration of the study
Who Masked: Outcomes Assessor
Masking Description: This is a pragmatic trial, so study participants and the investigator team will be unblinded to study procedures, however, the outcomes assessors (biostatistical team) will be blinded to arm assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: PharmFIT (Experimental): Subjects enrolled in the PharmFIT intervention will receive a referral notice from their primary care facility to pick up a FIT and receive support for screening from their pharmacist. After receiving the FIT and completing the FIT subject will receive their FIT results. Those with positive results will also be provided patient navigation support. This support will be provided by the pharmacist, in collaboration with the subject's PCP, and will include a) Discussing barriers to colonoscopy (e.g., fear, lack of transportation, inability to pay); b) Support for and confirmation of colonoscopy appointment scheduling; c) Review and support prep procedures; e) Post-procedure, discuss results and answer questions.
  Interventions: Behavioral: PharmFIT
- Control: Usual Care (No Intervention): Subjects randomized to this arm receive usual care.

INTERVENTIONS:
Behavioral: PharmFIT — The PharmFIT intervention involves the following components: referral notice to patient, FIT ready notification, FIT ready reminders, FIT distribution, FIT completion reminders, negative and positive results notification, patient navigation support.
  Arms: Intervention: PharmFIT

SUMMARY:
This study will conduct a randomized controlled trial to assess the impact of a pharmacy-based FIT intervention, Pharmacy-based FIT (PharmFIT), on colorectal cancer screening (CRC) screening rates in primary care patients who are not up to date on CRC screening. Through collaboration with community partners in North Carolina and the Pacific Northwest region, 1) the impact will be evaluated, 2) the implementation will be assessed, and 3) the costs of the PharmFIT intervention cost will be estimated. Patients (n=1,200) will be individually randomized to a usual care arm or a PharmFIT arm and we will determine whether there are statistically significant differences in CRC screening rates. Concurrently, a mixed methods approach will be used to assess a range of preliminary implementation outcomes, identify outcome barriers and facilitators, and identify implementation strategies to support future research. Also, the cost of PharmFIT will be calculated, using collaborative process flow diagramming (PFD) to inform micro-costing and budget impact analysis. Supported by preliminary work from the investigators, demonstrating widespread acceptability, feasibility, and preliminary effectiveness of PharmFIT, the rationale to conduct this hybrid 1 effectiveness-implementation trial1 is to generate new knowledge about pharmacy-based interventions to effectively increase CRC screening uptake and implementation. The central hypothesis is that the PharmFIT intervention will increase screening uptake by improving access to, and opportunities for, this preventive service through the involvement of a multidisciplinary, multisite, team-based care approach to CRC screening.

DETAILED DESCRIPTION:
The long-term goal of this study is to reduce CRC mortality by increasing access to CRC screening. The overall objective is to evaluate the effectiveness and implementation of a pharmacy-based FIT (PharmFIT) intervention. PharmFIT is a collaborative patient care service intervention that involves primary care clinics identifying active patients who are due for screening and referring them, outside of a medical visit, to community pharmacies to receive their CRC screening via FITs. The program consists of 1) Patient eligibility assessments and endorsement by the Primary Care Provider (PCP); 2) Counseling on FIT use and return by the pharmacists; 3) Reminders to complete screening by the pharmacy staff; 3) Test result communication by the pharmacists/PCPs; and 4) Patient navigation and care coordination for follow-up care by both pharmacists and PCPs.

ELIGIBILITY:
Inclusion Criteria: Clinic and pharmacy staff (n up to 100)

* Age ≥18 years
* Employed at a participating primary care clinic or pharmacy
* Fluent in English
* Has access to a computer with internet

Exclusion Criteria: Clinic and pharmacy staff

* Floaters/per diem employees
* Those who would object to having their interview audio recorded
* Those who would object to participation in evaluation surveys

Inclusion Criteria: Patients (n=1400)

* Age 45-75 years
* Patient at a participating primary care facility (medical visit within last 18 months)
* Current resident of NC or WA state
* Not up to date with recommended screening (e.g., no colonoscopy within 10 years, no FIT-DNA test within 3 years; no FIT/FOBT within 12 months)
* English and Spanish speakers
* Has access to a computer or smartphone with internet

Exclusion Criteria: Patients

* Previous USPST CRC screening within recommended screening period: 1) Colonoscopy within the past 10 years, 2) FIT/FOBT/FIT-DNA test within the past 12 months, 3) Previous sigmoidoscopy within the past 5 years, 4) Previous CT colonography within the past 10 years, 5) Other CRC screening tests
* CRC screening is contraindicated
* Previous positive FIT/FOBT/FIT-DNA
* Colorectal neoplasm or colorectal polyp
* Adenoma by biopsy
* Family history of colorectal cancer
* Diagnosed with inflammatory bowel disease
* Total or partial colectomy
* Diagnosis of Alzheimer's/other forms of severe dementia
* Resides in an assisted living facility
* Currently receiving hospice care
* Diagnosed with end stage renal disease
* Current diagnosis of certain cancers (e.g., CRC, mesothelioma, glioblastoma, lung, pancreatic, and liver/bile duct)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Service Penetration (Effectiveness) | 6-months post randomization
  Receipt of any USPSTF guideline recommended CRC screening (FIT, FIT-DNA, sigmoidoscopy, colonoscopy, CT colonography, or barium enema), using a yes ["1"] vs. no ["0"] dichotomous outcome in the 6 months following randomization.
Appropriateness of the PharmFIT intervention | 6-months post enrollment
  Perceptions that PharmFIT is agreeable, palatable, or satisfactory.
Acceptability of the PharmFIT intervention | 6-months post enrollment
  Perceptions that PharmFIT is relevant to, fits or is compatible with a given practice site, provider, or patient.
Feasibility of the PharmFIT intervention | 6-months post enrollment
  Extent to which PharmFIT was successfully implemented and used within the clinics and pharmacies, measured by the Implementation Outcomes Questionnaire (IOQ) Feasibility Subscale.
Fidelity to the PharmFIT intervention | Baseline, 6-months post enrollment
  PharmFIT delivered as intended; adherence; integrity; quality of PharmFIT intervention delivery, measured using the study's REDCap tracking database (e.g., patient communications delivered, FIT kits distributed, results reports, etc.).
Cost of the PharmFIT intervention | Through study completion, up to 12 months after PharmFIT intervention implementation
  Incremental cost of each additional patient screened in the intervention arm compared to usual care. Comparison of the programmatic costs incurred, and number of subjects screened in Arm 1(trial PharmFIT) compared to Arm 2 (usual care), measured as cost of intervention minus the cost of usual care, divided by the number screened in Arm 1 minus the number screened in Arm 2.
  Intervention costs will be assessed using periodic episodes of direct observation of PharmFIT outreach activities, time logs maintained by the intervention team, and assembly of administrative data capturing non-personnel/non-labor expenditures, such as costs associated with materials printing, FIT processing, and mailing costs. Usual care costs will be estimated using data collected from collaborative process flow diagramming sessions.

SECONDARY OUTCOMES:
Reach | 6-months post enrollment
  A) The total number of patients who received referrals after being identified for screening, overall and by patient sex, race, ethnicity, age group, insurance category, rurality, previous screening behavior, and clinic/pharmacy cluster. B) The number of patients who received referrals after being identified for screening, overall and by patient sex, race, ethnicity, age group, insurance category, rurality, previous screening behavior, and clinic/pharmacy cluster.
Timely FIT completion | 60 days post FIT receipt
  Proportion of patients randomized to PharmFIT who completed the FIT within 60 days.
Timely follow-up colonoscopy | 6-months post enrollment
  Proportion of patients with positive FIT results completing follow-up colonoscopy within 6 months following positive FIT results.

CONTACTS AND LOCATIONS:
Overall Officials: Alison T Brenner, PhD MPH, Principal Investigator — University of North Carolina, Chapel Hill; Parth D Shah, PharmD PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Fred Hutch Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data generated through this trial, including survey instruments and interview guides, will be made publicly available on the UNC Dataverse (https://dataverse.unc.edu/).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after trial results are published, or otherwise made available, with no end date.
Access Criteria: Deidentified trial data shared on the UNC Dataverse will be made publicly available without access criteria. Additional data or information may be made available upon request.
URL: https://dataverse.unc.edu/dataverse/cpcrn-4cnc-pharmfit

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials